CLINICAL TRIAL: NCT04375787
Title: High Dose Atorvastatin Raises Threshold of Contrast Induced Nephropathy in Diabetic Patients Undergoing Elective Coronary Intervention
Brief Title: Atorvastatin Effect on Contrast Induced Nephropathy in Diabetic Patients Undergoing Elective Coronary Intervention
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Mohamed Abdelfatah (Other)
Responsible Party: Sponsor-Investigator, Mohamed Abdelfatah, investigator, Assiut University
Organization: Assiut University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Atorvastatin in elective CA
Record Dates: First submitted 2020-05-04; First posted 2020-05-05 (Actual); Last update posted 2022-02-16 (Actual); Status verified 2022-02

CONDITIONS: Coronary Disease
MeSH Terms: conditions — Coronary Disease | interventions — Atorvastatin; Hydroxymethylglutaryl-CoA Reductase Inhibitors

STUDY DESIGN:
Intervention Model Description: 200 diabetic patients with indication for coronary intervention participated in the study. 100 patients were randomly assigned to receive atorvastatin (80 mg) just before coronary intervention (statin group) and 100 patients received placebo (control group).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Statin group (Active Comparator): 100 patients were randomly assigned to receive atorvastatin (80 mg) just before coronary intervention
  Interventions: Drug: Atorvastatin
- Placebo group (Placebo Comparator): 100 patients received placebo
  Interventions: Drug: Atorvastatin

INTERVENTIONS:
Drug: Atorvastatin — Patients received 80 mg atorvastatin before elective coronary angiography
  Other Names: statin

SUMMARY:
Investigate of the potential benefit of acute pretreatment with high dose atorvastatin (80 mg) in reduction of the incidence of CIN in diabetic patients indicated for elective coronary intervention.

DETAILED DESCRIPTION:
The study is a prospective, multi-center, randomized, placebo-controlled study. The ethical committee of the Faculty of Medicine, Assiut University approved the study protocol.

200 diabetic patients with indication for coronary intervention participated in the study. 100 patients were randomly assigned to receive atorvastatin (80 mg) just before coronary intervention (statin group) and 100 patients received placebo (control group). An informed written consent for participating in the study was obtained from each participant.

Exclusion criteria:

1. Current statin treatment within the previous three months.
2. Chronic renal failure patients on renal dialysis, or serum creatinine more than 1.5 mg/dl.
3. Severe co-morbidities i.e. patients with cancer, advanced liver cirrhosis.
4. Contraindications to statin therapy.
5. Contrast media injection within the preceding 10 days.
6. Pregnancy.
7. Refusal of consent. (B) Methodology:

All study patients were subjected to:

1. Full clinical history: including age, sex, history of smoking, hypertension, history of previous percutaneous coronary intervention (PCI), duration of diabetes mellitus (DM) and type of anti-DM treatment.
2. Thorough physical examination focusing on:

   * General examination including intra-procedural hemodynamic assessment.
   * Cardiac examination to elicit manifestations of heart failure.
3. Echocardiography searching for wall motion abnormalities and estimation of left ventricular systolic function.
4. Initial venous blood samples for determination of hemoglobin level and serum creatinine before the procedure. Follow up for serum creatinine at 48 hours post-procedure was done.

   CIN was stated as a raising of serum creatinine of more than 25% or ≥0.5 mg/dl (44 μmol/l) from initial level within 48 hours of the angiographic procedure and after excluding other factors that may cause nephropathy such as nephrotoxic drugs.
5. All patients received clopidogrel (600 mg) or ticagrelor (180 mg). Any nephrotoxic drugs (i.e., metformin, non-steroidal anti-inflammatory drugs) were withdrawn on admission.
6. Coronary intervention was done using the same non-ionic, low-osmolar contrast medium (Iopamidol; Scanlux, Sanochemia, Austria) in all cases.

   After the procedure, TIMI flow of the culprit artery was assessed, as well as the volume of used contrast media and time of X-ray exposure.
7. Statistical analysis:

Data were processed by statistical package for the social sciences (SPSS, version 20. 0). Descriptive statistics for interval and ordinal variables were calculated such as the ranges, means, and standard deviations, whereas, for categorical variables, the frequencies and percentages were reported. Student t-test or paired t-test, as appropriate, were used to compare normal and continuous variables. Chi-square test was used for comparing categorical variables. The level of significance was stated at P < 0.05. Receiver operating curves (ROC) were plotted and area under the curve (AUC) was assessed for some studied variables. Sensitivity and specificity were calculated at a cutoff point. A p value of <0.05 was considered significant.

ELIGIBILITY:
Inclusion Criteria:

* 200 diabetic patients with indication for coronary intervention participated in the study

Exclusion Criteria:

1. Current statin treatment within the previous three months.
2. Chronic renal failure patients on renal dialysis, or serum creatinine more than 1.5 mg/dl.
3. Severe co-morbidities i.e. patients with cancer, advanced liver cirrhosis.
4. Contraindications to statin therapy.
5. Contrast media injection within the preceding 10 days.
6. Pregnancy.
7. Refusal of consent.

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2020-03-15 (Actual); Primary Completion 2020-06-02 (Actual); Study Completion 2020-06-02 (Actual)

PRIMARY OUTCOMES:
Contrast Induced Nephropathy (CIN) | 48 hours
  CIN was defined as a rise of serum creatinine of more than 25% or ≥0.5 mg/dl (44 μmol/l) from baseline within 48 hours of the angiography

CONTACTS AND LOCATIONS:
Overall Officials: Ayman Ibrahem, MD, Study Chair — Assiut University; Ahmed Abdel-Galeel, MD, Study Director — Assiut University
Locations (1):
- Assiut University, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mohammed NM, Mahfouz A, Achkar K, Rafie IM, Hajar R. Contrast-induced Nephropathy. Heart Views. 2013 Jul;14(3):106-16. doi: 10.4103/1995-705X.125926. PMID 24696755
- [Background] Bolognese L, Falsini G, Schwenke C, Grotti S, Limbruno U, Liistro F, Carrera A, Angioli P, Picchi A, Ducci K, Pierli C. Impact of iso-osmolar versus low-osmolar contrast agents on contrast-induced nephropathy and tissue reperfusion in unselected patients with ST-segment elevation myocardial infarction undergoing primary percutaneous coronary intervention (from the Contrast Media and Nephrotoxicity Following Primary Angioplasty for Acute Myocardial Infarction [CONTRAST-AMI] Trial). Am J Cardiol. 2012 Jan 1;109(1):67-74. doi: 10.1016/j.amjcard.2011.08.006. Epub 2011 Sep 22. PMID 21943940
- [Background] Perrin T, Descombes E, Cook S. Contrast-induced nephropathy in invasive cardiology. Swiss Med Wkly. 2012 Jun 19;142:w13608. doi: 10.4414/smw.2012.13608. eCollection 2012. PMID 22714555
- [Background] McCullough PA, Adam A, Becker CR, Davidson C, Lameire N, Stacul F, Tumlin J; CIN Consensus Working Panel. Epidemiology and prognostic implications of contrast-induced nephropathy. Am J Cardiol. 2006 Sep 18;98(6A):5K-13K. doi: 10.1016/j.amjcard.2006.01.019. Epub 2006 Feb 10. PMID 16949375